CLINICAL TRIAL: NCT04852016
Title: Optimizing the Consent Process for Emergent Laparoscopic Cholecystectomy Using an Interactive Digital Education Platform: A Randomized Control Trial
Brief Title: Optimizing the Consent Process for Emergent Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Boris Zevin (Other)
Responsible Party: Sponsor-Investigator, Dr. Boris Zevin, Associate Professor of Surgery, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SURG-534-20
Record Dates: First submitted 2021-04-15; First posted 2021-04-21 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Consent; Laparoscopic; Cholecystectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Educational Platform (Experimental): Study participants randomized to the DEP+SVC group (intervention) will be presented with an iPad with a link to an interactive DEP module discussing the indications for LC, alternatives, risks, complications, expectations and anticipated recovery. They will be asked to review the DEP module at their own pace and will be required to confirm understanding of all of the material presented on the DEP. Upon completion of the module, a member of the surgery team will ask the patient if they have any additional questions or require further clarification regarding the LC procedure, indications for surgery, alternatives, risk, complications, expectations and anticipated recovery. Once all of participant's questions are answered, an informed paper-based consent form for LC will be signed.
  Interventions: Behavioral: Consent process with the addition of Digital educational platform (DEP)
- Standard Verbal Consent (Active Comparator): Study participants randomized to the SVC group (control) will discuss the LC procedure, indications for surgery, alternatives, risk, complications, expectations and anticipated recovery with a member of the surgery team. The study participant will be given the opportunity to ask questions and once all of the questions have been answered, an informed paper-based consent form for LC will be signed.
  Interventions: Behavioral: Consent process using the standard verbal consent (SVC)

INTERVENTIONS:
Behavioral: Consent process with the addition of Digital educational platform (DEP) — In-patients being consented for laparoscopic cholecystectomy will be provided with a Digital Educational Platform (DEP), in the form of modules on an iPad. These participants will still undergo the usual standard verbal consent (SVC). Multiple choice questionnaires will be given pre and post consent to determine acquisition and retention of the information provided using DEP.
  Arms: Digital Educational Platform
Behavioral: Consent process using the standard verbal consent (SVC) — In-patients being consented for laparoscopic cholecystectomy will go through the SVC. Multiple choice questionnaires will be given pre and post consent to determine acquisition and retention of the information provided using SVC.
  Arms: Standard Verbal Consent

SUMMARY:
The Canadian Medical Protective Association (CMPA) defines informed consent (IC) as a voluntary process where important elements include details of the procedure, complications, and proposed alternatives. Laparoscopic cholecystectomy (LC) was the most common laparoscopic procedure cited in 423 medical-legal cases reported by CMPA in 2017, with 29% of cases citing issues in pre-operative care including inadequacy of the consent process. The investigators recently demonstrated that technology can help improve the IC process in an outpatient setting by conducting a prospective randomized controlled trial to examine the effects of adding a digital educational platform (DEP) module to a standard verbal consent (SVC) for an elective laparoscopic Roux-en-Y gastric bypass procedure. The investigators demonstrated a significant improvement in immediate post-consent knowledge of the risks, benefits and alternatives in patients who viewed the DEP module with equivalent patient satisfaction as compared to a SVC. With the proposed study the investigators plan to gather evidence to support implementing a digital education platform for emergent surgical procedures performed in an in-patient setting.

The investigators propose to conduct a randomized controlled trial to explore the benefits of adding a DEP module to a SVC for patients presenting with acute cholecystitis requiring an emergent LC as an in-patient. Participants will be randomly allocated (1:1) to either a control group (SVC) or an intervention group (SVC + DEP). Primary outcome of interest will be immediate post-consent knowledge of the risks, benefits, alternatives and expected outcomes for a LC. Secondary outcomes will include satisfaction with the consent discussion and delayed retention of knowledge of the risks, benefits, alternatives and expected outcomes for a LC .

The investigators hypothesize that completion of the DEP module in addition to SVC will result in superior immediate and delayed post-consent knowledge of risks and benefits of LC with equivalent patients satisfaction as compared to SVC alone.

The results of this study will provide evidence supporting the addition of DEP to SVC for urgent and emergent surgical procedures.

DETAILED DESCRIPTION:
Required elements for an informed consent (IC) in surgery have been well established. The Canadian Medical Protective Association (CMPA) defines IC as a voluntary process where important elements include details of the procedure, complications, and proposed alternatives. The individual should also be given ample time to ask questions to ensure best understanding of the procedure. Shortcomings in the process can lead to patient complaints, unmet expectations and have significant legal ramifications. Of all medical-legal cases involving inadequacy of informed consent reported by CMPA in 2016, 65% involved surgical procedures and 79% had unfavorable outcomes. Laparoscopic cholecystectomy (LC) was the most common laparoscopic procedure cited in 423 medical-legal cases reported by CMPA in 2017, with 29% of cases citing issues in pre-operative care including inadequacy of the informed consent process.

The investigators conducted a retrospective chart review of 270 patients who underwent 71(26%) elective and 199(74%) emergent LC at our tertiary academic centre and demonstrated poor documentation of IC with only 5(2%) patients' charts having complete documentation of all three elements of IC. For emergent cases, discussion of possible complications of LC was documented 174(64%) of cases; details of the LC were documented in 7(2.6%) of cases; and alternatives to LC were documented in 3(1.1%) of cases. Emergent LC was associated with worse documentation of IC as compared to elective LC. It is difficult to ascertain whether poor documentation is associated with poor informed consent discussions; however, use of digital education platforms (DEP) can enhance a patient's understanding of the risks, benefits and alternatives to a proposed operative procedure and can ensure the comprehensiveness of the consent discussion.

The investigators recently conducted a prospective randomized controlled trial of 51 patients with severe obesity to examine the effects of adding a digital educational platform (DEP) to a standard verbal consent (SVC) for a laparoscopic Roux-en-Y gastric bypass procedure. In this study the investigators demonstrated that addition of DEP to SVC resulted in improved knowledge of the risks, benefits and alternatives to the procedure vs SVC alone (85.0±8.8% vs 78.7±8.7%; p=0.01; Effect Size=0.72), equivalent patient satisfaction (31.5±1.1 vs 31±2.7; p=0.10), and significantly shorter face-to-face time between patient and surgeon to obtain informed consent (358±198sec vs 751±212sec; p<0.01; Effect Size=1.92). However, the generalizability and transferability of our findings to an inpatient setting and to emergent operations is currently unknown.

The investigators will be conducting a randomized controlled trial to explore the benefits of adding a DEP module to a SVC for patients presenting with acute biliary pathology requiring an emergent LC in an in-patient setting.

Significance:

Although addition of the DEP to SVC has been shown to result in improved patient understanding of risks, benefits and alternatives of a proposed operation in an elective setting, there is a paucity of data in an emergent acute care setting where the environment can be chaotic with shortened time for comprehensive informed consent discussions. The investigators hope that the results of this study will not only provide the evidence to support adding DEP to SVC for emergent surgical procedures, but will also improve informed consent discussions and patients' comprehension of the risks and benefits of proposed procedures in an acute care setting.

Hypotheses:

1. Participants in the intervention (DEP + SVC) group will demonstrate greater immediate and delayed (4-6 weeks) post-consent knowledge of the risks, benefits, alternatives and expected outcomes for the LC operation as compared to participants in the control (SVC) group.
2. Participants in the intervention (DEP + SVC) group will demonstrate equivalent satisfaction with the consent process as compared to participants in the control (SVC) group.

Methods:

Study Design and Setting:

This study will be a prospective non-blinded randomized control trial conducted at Kingston Health Sciences Centre (tertiary academic hospital in Kingston, Ontario, Canada). The investigators will recruit patients who are admitted to hospital with biliary pathology to undergo an emergent laparoscopic cholecystectomy (LC). Study participants will be randomly allocated in a 1:1 ratio to a control group (SVC) or an intervention group (DEP+SVC).

Recruitment and Randomization:

Patients (potential study participants) will be invited to participate in the current study once a clinical decision to recommend laparoscopic cholecystectomy has been made. Randomization will occur 1:1 to either an intervention (DEP+SVC) or a control group (SVC) using a sealed envelope technique.

Baseline Data:

The investigators will use the online Qualtrics platform to collect all of the demographic and outcomes data for this study. For baseline data, the investigators will collect participant data including age, sex, level of education ("did not complete high school", "high school", "college", "university"), background in a medical field (yes/no), previous consultation with a surgeon regarding laparoscopic cholecystectomy (yes/no). The investigators will also document the setting in which the consent discussion took place (emergency room or surgery ward), as well as admission diagnosis (biliary colic, acute cholecystitis, gallstone pancreatitis, choledocholithiasis, cholangitis) (Appendix 1) The investigators will ask study participants to complete a baseline basic English literacy reading test (Appendix 2), a self-reported rating of their understanding of the LC operation (scale of 1 to 10), and a multiple-choice knowledge test (MCQ, 20 questions, maximum score 20) assessing baseline knowledge of LC, indications for surgery, alternatives, risk, complications, and anticipated recovery. The knowledge test will be piloted with relevant stakeholders including general surgeons and patients who have undergone a LC prior to its use in the study. Participants will not be made aware of the correct answers to the questions on the test.

Standard Verbal Consent (control group):

Study participants who are randomized to the control (SVC) group will discuss the LC procedure, indications for surgery, alternatives, risks, complications, expectations and anticipated recovery with a member of the surgery team. The study participant will be given the opportunity to ask questions and once all of the questions have been answered, a standard informed consent form for LC will be signed.

Digital Education Platform (intervention group):

Study participants who are randomized to the intervention (DEP+SVC) group will be presented with an iPad an interactive DEP module discussing the indications for LC, alternatives, risks, complications, expectations and anticipated recovery. Participants will be asked to review the DEP module at their own pace and will be required to confirm understanding of all of the material presented on the DEP. They will have the opportunity to move back and forth within the module until they are satisfied. Upon completion of the module, a member of the surgery team will ask the patient if they have any additional questions or require further clarification regarding the LC procedure, indications for surgery, alternatives, risks, complications, expectations and anticipated recovery. Once all of participant's questions are answered, a standard informed consent form for LC will be signed.

Primary Outcome:

Knowledge of LC procedure, indications for surgery, alternatives, risks, complications, expectations and anticipated recovery will be measured using the same knowledge test (20 questions, maximum score 20) as for baseline knowledge assessment. The knowledge test will be completed right after the informed consent form is signed for LC.

Secondary Outcomes:

Self-reported understanding of the LC operation after signing of the informed consent will be assessed by asking study participants to rate their understanding on a scale of 1 to 10. Retention of knowledge about the LC procedure, indications for surgery, alternatives, risks, complications, expectations and anticipated recovery will be assessed in 4-6 weeks using the same knowledge test (20 MCQ questions, maximum score 20) as for baseline assessment. This delayed knowledge test will be administered on the day of patient's follow-up appointment with the surgeon, which is usually 4-6 weeks after their discharge from hospital.

Participant's satisfaction with the clinical encounter will be assessed using a modified Client Satisfaction Questionnaire (CSQ-8, maximum score 32) - a validated assessment tool of patient satisfaction[6] - at the end of the consent discussion after signing the informed consent form for LC (Appendix 3).

Sample Size:

Based on the results from the investigator's previous study, assuming a standard deviation of 9.0 and medium Cohen's d effect size of 0.66 for the MCQ knowledge test, the investigators will plan to recruit 36 patients per group to detect a 1.2 point difference in MCQ score (6%) change between two groups, with 80% power for the two sample t test (α = 0.05).

Statistical Analysis:

Demographic data will be compared between groups using the Student's t test (continuous variables) and Chi squared test (categorical variables). Participant satisfaction scores and knowledge test scores will be compared between groups using a Student's t test. Within group changes (eg. baseline vs immediate post test) in knowledge test scores with be compared using a paired t-test. Effect sizes will be calculated using Cohen's d. Statistical significance will be set to α = 0.05.

Timeline:

March 2021-May 2021:

Pilot testing of knowledge MCQ with key stakeholders (surgeons and patients) Creation of the DEP module for laparoscopic cholecystectomy Creation of online data collection forms (baseline testing and post-intervention testing) using Qualtrics

June 2021 - February 2023 Participant recruitment, randomization and data collection

January 2023 - February 2023 Data analysis Manuscript and abstract preparation

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older
* Individuals admitted to Kingston Health Sciences Centre with acute cholecystitis
* Must be able to read, write and speak English
* Must be able to provide consent

Exclusion Criteria:

* Individuals who are not able to provide informed consent for laparoscopic cholecystectomy.
* Individuals who are not able to access and view the interactive digital education platform
* Individuals who can not read, write or speak English

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Knowledge of the Laparoscopic Cholecystectomy Procedure | 1 day
  Understanding indications for surgery, alternatives, risks, complications, expectations and anticipated recovery will be one of the primary outcomes for this study. A 20 question multiple choice questionnaire will be used to measure this outcome.

SECONDARY OUTCOMES:
Self-reported rating of understanding of the laparoscopic cholecystectomy procedure. | 1 day
  Participants will be asked to rate their understanding of the procedure on a scale from 0-10 (0 - no prior knowledge/10 - I know everything).
Retention of Knowledge | 4-6 weeks
  Participants will complete a 20 question multiple choice test 4-6 weeks after their operation (during their follow up appointment).
Participant satisfaction with the clinical encounter | 1 day
  Participant satisfaction will be assessed using a modified Client Satisfaction Questionnaire (CSQ-8, maximum score 32) at the end of the consent discussion.

CONTACTS AND LOCATIONS:
Overall Officials: Boris Zevin, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zevin B, Almakky M, Mancini U, Robertson DI. Digital approach to informed consent in bariatric surgery: a randomized controlled trial. Surg Endosc. 2022 Jan;36(1):809-816. doi: 10.1007/s00464-020-08277-x. Epub 2021 Jan 27. PMID 33502615